CLINICAL TRIAL: NCT07070037
Title: Five-Year Visual Function and Refractive Outcomes After Congenital Cataract Surgery: A Multicenter Observational Cohort Study
Brief Title: Five-Year Visual Function and Refractive Outcomes After Congenital Cataract Surgery
Status: Recruiting | Type: Observational
Sponsor: Jin Yang (Other)
Responsible Party: Sponsor-Investigator, Jin Yang, Chief Physician, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Other Study IDs: Congenital Cataract-2025-001
Record Dates: First submitted 2025-06-29; First posted 2025-07-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-06

CONDITIONS: Congenital Cataract; Pediatric Cataract
Keywords: Congenital Cataract; Pediatric Cataract Surgery; Visual Function; Stereopsis; Amblyopia; Long-term Outcomes
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- congenital cataract: congenital cataract

SUMMARY:
This prospective multicenter observational study aims to evaluate the 5-year visual function and refractive outcomes in children undergoing surgery for congenital cataract. Key outcomes include best-corrected visual acuity, stereopsis, refractive error, and axial length growth. The study will help identify long-term trends and prognostic indicators after early cataract intervention in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital cataract
* Underwent cataract extraction before 1 year of age
* Available for regular follow-up for at least 5 years postoperatively
* Written informed consent from legal guardian

Exclusion Criteria:

* Acquired cataract or traumatic origin
* Associated ocular malformations (e.g., microphthalmia, coloboma)
* Systemic syndromes affecting vision (e.g., Down syndrome)
* History of secondary surgery affecting visual outcome

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll pediatric patients diagnosed with congenital cataract who underwent cataract extraction with or without intraocular lens (IOL) implantation. Participants must be able to complete regular postoperative follow-up assessments from the time of surgery up to 5 years. Both unilateral and bilateral cases are eligible. The study population is recruited from multiple tertiary eye centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  UDVA and BCVA will be assessed using age-appropriate optotypes (e.g., Snellen chart, ETDRS chart, or Lea symbols) and recorded in logMAR units at the last available follow-up, with a minimum duration of 5 years postoperatively.
axial length | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  AL
Refractive Error | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  Refractive Error

SECONDARY OUTCOMES:
IOP | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  intraocular pressure
Corneal Curvature (K1 and K2) by Pentacam | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  Flat (K1) and steep (K2) corneal curvature values will be measured using Pentacam and recorded in diopters (D).
Stereopsis | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  Stereopsis will be assessed using age-appropriate tools (e.g., Randot Preschool or Titmus Fly Test) and reported in seconds of arc. Loss of stereopsis is defined as >3000 arcsec.
white to white | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  WTW (mm)
anterior chamber depth | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  ACD(mm)
Complications | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  Any postoperative complications following congenital cataract surgery, including glaucoma, anterior capsular opacification (ACO), etc.
Central Corneal Thickness (CCT) | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  Corneal pachymetry will be measured with Pentacam at the central point and reported in microns (µm).
Corneal Astigmatism Magnitude | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  Corneal astigmatism will be calculated from the difference between steep and flat meridians (K2-K1) using Pentacam data, and reported in diopters.
Binocular Fusion Assessment | Participants will be followed at 1 week, 1 month, 3 months, 6 months, and annually from 1 to 5 years postoperatively.
  Binocular fusion will be evaluated using the Worth 4-Dot test under near and distance conditions. Results will be categorized as "fusion", "suppression", or "alternation".

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Study Chair — Fudan University
Locations (1):
- Eye and ENT hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No